CLINICAL TRIAL: NCT05312411
Title: A Phase I Feasibility And Safety Study of Fluorescein-Specific (FITC-Ew) CAR T Cells In Combination With Parenterally Administered Folate-Fluorescein (UB-TT170) For Osteogenic Sarcoma
Brief Title: A Phase I Feasibility And Safety Study of Fluorescein-Specific (FITC-E2) CAR T Cells In Combination With Parenterally Administered Folate-Fluorescein (UB-TT170) For Osteogenic Sarcoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Umoja Biopharma (Industry)
Responsible Party: Principal Investigator, Colleen Annesley, Medical Director, Seattle Children's Therapeutics, Seattle Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENLIGHTen-01
Record Dates: First submitted 2019-03-20; First posted 2022-04-05 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Osteosarcoma
Keywords: osteosarcoma; bone cancer; pediatric sarcoma; young adult sarcoma
MeSH Terms: conditions — Osteosarcoma; Bone Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- UB-TT170 following SCRI-E2CAR_EGFrtv1 (Experimental): Following CAR T cell administration, subjects will receive a first Course of 3 escalating doses of UB-TT170 over 2 weeks followed by fixed weekly dosing for 2 weeks. If eligible, subjects may proceed to Courses 2 - 4 consisting of 7 weekly doses of UB-TT170.
  Interventions: Biological: SCRI-E2CAR_EGFRtv1; Drug: UB_TT170

INTERVENTIONS:
Biological: SCRI-E2CAR_EGFRtv1 — Autologous CD4+ and CD8+ T cells that have been genetically modified to express antiFL(FITC-E2)
Drug: UB_TT170 — Bispecific small molecule adapter formulated with phosphate buffered saline

SUMMARY:
The purpose of this study is to see if a new treatment could help patients who have osteosarcoma that does not go away with treatment (is refractory) or comes back after treatment (is recurrent).This study is testing a combination of study therapies, UB-TT170 and genetically modified chimeric antigen receptor T lymphocyte (CAR T) cells, which work together in a way that is different from chemotherapy.

In this study, researchers will take some of your blood and remove the T cells in a process called "apheresis". Then the T cells are taken to a lab and changed to CAR T cells that recognize the flags from UB-TT170. Once researchers think they have grown enough CAR T cells, called antiFL(FITC-E2) CAR T cells, to fight your cancer, you may get some chemotherapy to make room in your body for the new cells and then have those cells put back in your body.

A few days after the you get your CAR T cell infusion you will start to get infusions of UB-TT170, with the dose slowly increasing for the first few infusions until you have reached a maximum dose that you will get on a regular schedule. The UB-TT170 will attach to your tumor cells and flag them so that they attract the CAR T cells. When the CAR T cells see the labeled tumor cells they can kill the tumor cells.

The active part of the study lasts about 8 months, and if you get the CAR T cell infusion you will be in long-term follow-up for 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Refractory or recurrent/progressive osteosarcoma that has failed first line therapy for Osteosarcoma per NCCN or upfront Children's Oncology Group clinical trial and is not amenable to surgical resection (must meet one of the following):

  1. New site of measurable disease by radiographic imaging or histologic confirmation
  2. New site of evaluable disease by radiographic imaging (including FDG-PET) or histologic confirmation
  3. Greater than 20% increase in at least one tumor dimension documented by CT/MRI, AND a maximum absolute increase of 5 mm in longest dimension of existing lesion(s) (previously irradiated lesions may be included)
  4. Persistent measurable disease or FDG-PET avid bone metastasis that has failed to achieve complete remission to upfront conventional therapy (surgery, radiotherapy and/or chemotherapy)
* Able to tolerate apheresis, including placement of temporary apheresis catheter, if necessary, or already has an apheresis product available for use in manufacturing
* Life expectancy ≥ 8 weeks
* Lansky or Karnofsky score ≥ 50
* Anti-cancer agents, radiotherapy, cytoxic chemotherapy, biologic therapy, anti-tumor antibody therapy, genetically modified cell therapy, and, if no apheresis product available, corticosteroid therapy (excluding physiologic replacement), discontinued within protocol specified wash-out period
* Adequate hematologic, renal, hepatic, cardiac, and respiratory function.
* Negative HIV, hepatitis B and C test within 3 months
* If of child-bearing or fathering potential, willing to use highly effective contraception through 12 months following final stud drug infusion

Exclusion Criteria:

* Active malignancy other than primary malignant solid tumor diagnosis (CNS intracranial metastases are allowed)
* Ongoing, symptomatic CNS pathology requiring medical intervention
* Receiving external beam radiotherapy
* Presence of active, severe infection
* Primary immunodeficiency syndrome
* Pregnant or breast feeding
* Unwilling to provide consent/assent for study participation, including 15 year follow up
* Presence of any condition that, in the opinion of the investigator, would prohibit the subject from undergoing treatment under this protocol.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2040-05 (Estimated)

PRIMARY OUTCOMES:
Adverse events associated with ex-vivo expanded autologous T cells genetically modified to express an antiFL(FITC-E2) CAR administered with UB-TT170 will be assessed | 30 days
  The type, frequency, severity, and duration of adverse events will be summarized

SECONDARY OUTCOMES:
Ability to manufacture antiFL(FITC-E2) CAR cells | 28 Days
  The number of successfully manufactured antiFL(FITC-E2) CAR products will be assessed
Evaluate the pharmacokinetics of UB-TT170 in combination with the anti-FL(FITC-E2) CAR T cells | 25 days
  Pharmacokinetics of UB-TT170 in combination with the anti-FL(FITC-E2) CAR T cells

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Albert, MD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No